CLINICAL TRIAL: NCT06911489
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Tolerability of 68Ga-NRT6020 Injection and 177Lu-NRT6020 Injection in FAP-Positive Participants With Advanced Solid Tumors
Brief Title: Safety Trial of 68Ga/177Lu-NRT6020 in FAP-Positive Advanced Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu New Radiomedicine Technology Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NRT6020-101
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Malignancy
Keywords: solid tumor; Radionuclide Drug Conjugates; Companion Diagnostics; FAP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 68Ga-NRT6020 Injection (stage 1) (Experimental): Stage 1 is designed as a single-arm, single-dose study, planning to enroll participants with advanced solid tumors, with two planned dose groups: a low-dose group and a high-dose group. The dose groups are sequentially enrolled from low to high, with 6 participants planned for enrollment in each dose group.
  Interventions: Diagnostic Test: 68Ga-NRT6020 Injection
- 68Ga-NRT6020 Injection+ 177Lu-NRT6020 Injection (stage 2) (Experimental): Stage 2 is designed as a single-arm, multiple-dose, "3+3" dose-escalation study, and will enroll FAP-positive patients with advanced solid tumors who have failed or have no available standard therapy.
  Interventions: Diagnostic Test: 68Ga-NRT6020 Injection; Drug: 177Lu-NRT6020 Injection (stage 2)
- 68Ga-NRT6020 Injection+ 177Lu-NRT6020 Injection (stage 3) (Experimental): This stage 3 of the study is designed as a multi-center, single-arm, multiple-dose, parallel-cohort study, and will enroll FAP-positive patients with advanced solid tumors who have failed or have no available standard therapy.
  Interventions: Diagnostic Test: 68Ga-NRT6020 Injection; Drug: 177Lu-NRT6020 Injection (stage 3)

INTERVENTIONS:
Diagnostic Test: 68Ga-NRT6020 Injection — Participants will receive a single intravenous injection of 68Ga-NRT6020 Injection (3 mCi or 5 mCi) and PET/CT scans at multiple time points.
Drug: 177Lu-NRT6020 Injection (stage 2) — It is planned to evaluate 4 dose levels of 177Lu-NRT6020 Injection: 50mCi, 100mCi, 150mCi and one/more adaptive dose groups (ranged from 150 to 250 mCi, the specific doses and/or doses with other frequencies within the range of 150~250mCi, need to be determined after the completion of the dose-limiting toxicity (DLT) assessment for the previous three dose groups, in combination with the safety, pharmacokinetics and radiation dosimetry results of the participants, following confirmation by the SRC) which will be administered every 6 weeks (Q6W), and/or other dosing intervals determined by the SRC, for up to 6 cycles.
  Arms: 68Ga-NRT6020 Injection+ 177Lu-NRT6020 Injection (stage 2)
Drug: 177Lu-NRT6020 Injection (stage 3) — Participants will receive intravenous injection of 177Lu-NRT6020 Injection, administered Q6W and/or other dosing intervals determined by the SRC, for up to 6 cycles.
  Arms: 68Ga-NRT6020 Injection+ 177Lu-NRT6020 Injection (stage 3)

SUMMARY:
Stage 1 (Safety study for 68Ga-NRT6020 Injection):

The goal of this clinical trial stage is to evaluate the safety of 68Ga-NRT6020 Injection in participants with advanced solid tumors. The study will also assess the biodistribution, radiation dosimetry, imaging profile, and pharmacokinetics of the drug. Additionally, researchers aim to investigate how consistent the PET/CT imaging results of 68Ga-NRT6020 are with 18F-FDG PET/CT imaging and FAP immunohistochemistry (IHC) results.

Stage 2 (Safety and tolerability study for 177Lu-NRT6020 Injection):

This stage focuses on evaluating the safety and tolerability of 177Lu-NRT6020 Injection in FAP-positive participants with advanced solid tumors. Researchers will also assess the safety of 68Ga-NRT6020 Injection in this population. The study will evaluate the biodistribution, radiation dosimetry, pharmacokinetics, and preliminary efficacy of 177Lu-NRT6020 Injection. Additionally, the imaging profile of 68Ga-NRT6020 and its consistency with other imaging techniques will be further investigated.

Stage 3 (Preliminary efficacy study for 68Ga/177Lu-NRT6020 Injection):

The objective of this stage is to evaluate the safety of 177Lu-NRT6020 Injection and 68Ga-NRT6020 Injection in FAP-positive participants with advanced solid tumors, as well as to determine the recommended phase 2 dose (RP2D) of 177Lu-NRT6020 Injection. The study will also assess the preliminary efficacy, biodistribution, radiation dosimetry, and pharmacokinetics of the drugs. Furthermore, researchers will investigate the imaging profile of 68Ga-NRT6020 and its consistency with other imaging techniques.

DETAILED DESCRIPTION:
During the study, 68Ga-NRT6020 served as the companion diagnostic agent for 177Lu-NRT6020 to select eligible patients. This stage 2 and stage 3 of the study is designed as a multi-center, multiple-dose, parallel-cohort study, and will enroll FAP-positive (FAP-positive is defined by positive PET/CT imaging results for 68Ga-NRT6020; and dose of 68Ga-NRT6020 will be confirmed by the SRC after stage 1) patients with advanced solid tumors who have failed or have no available standard therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants aged 18-80;
2. Histologically or cytologically confirmed advanced solid tumors; advanced solid tumors patients who have failed prior standard therapies or deemed unsuitable for standard therapies (only for stage 2 and stage 3);
3. Have at least one measurable lesion as per RECIST v1.1/PERCIST criteria;
4. For stage 2 and stage 3, a positive 68Ga-NRT6020 Injection PET/CT imaging results is required;
5. Participants must have adequate organ function;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy ≥3 months;
8. For women of childbearing potential, a negative blood pregnancy test within 3 days before the first dose is required, and fertile male and female participants of childbearing potential must agree to use effective contraception with their partners from the signing of the informed consent form until 12 months after the last dose of the investigational drug.

Key Exclusion Criteria:

1. Known allergy to 68Ga-NRT6020 Injection, 177Lu-NRT6020 Injection, or any of their ingredients, such as alcohol;
2. Presence or suspicion of primary central nervous system tumors or intracranial metastasis;
3. For stage 1: Received prior antitumor treatments within 7 days before the investigational drug dosing, and/or plan to receive antitumor treatments during the safety observation period; For stage 2 and stage 3: Received prior antitumor treatments within 4 weeks before the initial investigational drug dosing, including chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc.;
4. History of other malignancies within 5 years prior to the first dose of the investigational drug, excluding cured non-melanoma skin cancer, early-stage papillary thyroid cancer, and cervical carcinoma in situ;
5. Presence of severe or uncontrolled cardiac diseases requiring treatment;
6. High risk of bleeding;
7. Active syphilis or human immunodeficiency virus (HIV) antibody positive;
8. HBsAg-positive or HBcAb-positive with HBV-DNA levels above the detection limit;
9. Failure to alleviate previous antitumor treatment toxicities to Grade 0 or 1 according to CTCAE v5.0;
10. Participate in any other clinical trials within 1 month before the first dosing of 68Ga-NRT6020 Injection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 1 year
  Occurrence of adverse events
Dose-limiting toxicity (DLT) (stage 2) | After the first dose of 177Lu-NRT6020 administration, up to 42 days
  Evaluate the safety and tolerability of 177Lu-NRT6020
Maximum tolerated dose (MTD) (if any) or recommended dose for expansion study of 177Lu-NRT6020 Injection (stage 2) | Through study completion, an average of 1 year
  Evaluating the safety and tolerability of 177Lu-NRT6020 with the aim of determining the optimal dose
RP2D for 177Lu-NRT6020 Injection (stage 3) | Through study completion, an average of 1 year
  Determine the optimal dose of 177Lu-NRT6020

SECONDARY OUTCOMES:
Standardized uptake values (SUV) (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Evaluate the distribution of 68Ga-NRT6020 Injection in various tissues and organs of the human body
Absorbed dose (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Evaluate the dosimetry characteristics of 68Ga-NRT6020 Injection in various tissues and organs of the human body
Effective dose (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Evaluate the dosimetry characteristics of 68Ga-NRT6020 Injection in the human body
Scanning time window (stage 1) | After the administration of 68Ga-NRT6020, within 3 hours
  Compare the imaging parameter in different timepoints and different doses
Radioactivity in biological specimen (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Detect the radioactivity in specimen samples at various time points
Peak Plasma Concentration (Cmax) of 68Ga-NRT6020 (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Time to reach maximum concentration (Tmax) of 68Ga-NRT6020 (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Area under the plasma concentration versus time curve (AUC) of 68Ga-NRT6020 Injection (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Half life (t1/2) of 68Ga-NRT6020 (stage 1) | After the administration of 68Ga-NRT6020, within 24 hours
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Standardized uptake values (SUV) (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Evaluate the distribution of 177Lu-NRT6020 Injection in various tissues and organs of the human body
Absorbed dose (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Evaluate the dosimetry characteristics of 177Lu-NRT6020 Injection in various tissues and organs of the human body
Effective dose (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Evaluate the dosimetry characteristics of 177Lu-NRT6020 Injection in the human body
Objective response rate (ORR) (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the investigator in accordance with the RECIST v1.1/PERCIST criteria
Duration of response (DOR) (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the investigator in accordance with the RECIST v1.1/PERCIST criteria
Progression-free survival (PFS) (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the investigator in accordance with the RECIST v1.1/PERCIST criteria
Radioactivity in biological specimen (stage 2) | After the administration of 177Lu-NRT6020, at least 7 days
  Detect the radioactivity in specimen samples at various time points
Peak Plasma Concentration (Cmax) of 177Lu-NRT6020 (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Time to reach maximum concentration (Tmax) of 177Lu-NRT6020 (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Area under the plasma concentration versus time curve (AUC) of 177Lu-NRT6020 (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Half life (t1/2) of 177Lu-NRT6020 (stage 2 and stage 3) | After the administration of 177Lu-NRT6020, at least 7 days
  Multiple blood samples will be collected to determine the pharmacokinetic profiles of 68Ga-NRT6020 Injection
Objective response rate (ORR) (stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the Independent Review Committee (IRC) in accordance with the RECIST v1.1/PERCIST criteria
Duration of response (DOR) (stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the Independent Review Committee (IRC) in accordance with the RECIST v1.1/PERCIST criteria
Progression-free survival (PFS) (stage 3) | After the administration of 177Lu-NRT6020, within 1 year
  Evaluated by the Independent Review Committee (IRC) in accordance with the RECIST v1.1/PERCIST criteria

OTHER OUTCOMES:
Consistency of 68Ga-NRT6020 Injection PET/CT imaging | After the administration of 68Ga-NRT6020, within 3 hours
  Evaluate the consistency between 68Ga-NRT6020 Injection PET/CT imaging and 18F-FDG PET/CT imaging results, as well as the consistency of 68Ga-NRT6020 Injection PET/CT imaging with FAP IHC results.
Scanning time window (stage 2) | After the administration of 68Ga-NRT6020, within 3 hours
  Compare the imaging parameter in different timepoints and different doses
Imaging dose of 68Ga-NRT6020 Injection (stage 3) | After the administration of 68Ga-NRT6020, within 3 hours
  Compare the imaging parameter under different doses in order to select the optimal imaging dose
Scanning time window (stage 3) | After the administration of 68Ga-NRT6020, within 3 hours
  Compare the imaging parameter in different timepoints and different doses

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Insititute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No